CLINICAL TRIAL: NCT04934865
Title: Real Life Prospective Multicentric Study Evaluating the Clinical and Organisational Impact of Moovcare® Lung Connected Medical Device in Lung Cancer Patients : REAL-MOOV-LUNG
Brief Title: Real Life Study Evaluating the Clinical and Organisational Impact of Moovcare® Lung Connected Medical Device in Lung Cancer Patients : REAL-MOOV-LUNG
Acronym: REAL-MOOV-LUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2020-13
Record Dates: First submitted 2021-06-08; First posted 2021-06-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated for their lung cancer and Moovcare® Lung follow-up. (Other)
  Interventions: Device: Patients treated for their lung cancer.

INTERVENTIONS:
Device: Patients treated for their lung cancer. — In addition to the weekly Moovcare® Lung follow-up, patients will benefit from standard oncological follow-up at the discretion of their oncologist according to standard recommendations for 2 years. Questionnaires will be completed at different times as mentioned below on the global study scheme and Flowchart.
  In an active treatment situation, the pace of consultations will be adapted to the pace of treatment administration, according to standard recommendations. It may be lengthened in the absence of a clinical application or biological alert at the discretion of the investigator.

SUMMARY:
Evaluation of patient's proportion, whose management care has been modified at least once and specially by Moovcare® Lung application at 12 and 24 months.

DETAILED DESCRIPTION:
Primary objective of the study:

The primary objective is a clinical one and is to evaluate the proportion of patients, whose management care has been modified at least once and specially by Moovcare® Lung application at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with lung cancer at any diagnostic stage and histology.
2. Patient willing to use the follow-up setting with Moovcare® Lung apps.
3. Age ≥ 18 years.
4. Patient received anti-cancer treatment (surgery, chemotherapy, radiation (stereotaxy or not) or radio-chemotherapy association ended less than 12 weeks (Cohort 1 post-treatment); or during maintenance treatment or consolidation by chemotherapy or targeted therapy, or by immunotherapy initiated less than 12 weeks (Cohort 2 during treatment).
5. Imaging tumor evaluation less than 12 weeks showing disease control (response or stability according to RECIST 1.1 criteria).
6. Patient with symptomatic score on Moovcare® Lung apps less than 7.
7. Patient (or relatives) with internet access, a personnal e-mail box and a smartphone.
8. Patient with social security affiliation.
9. Signed informed consent form.

Exclusion Criteria:

1. Patient with progression after the first evaluation of initial treatment.
2. Pregnancy and breast-feeding.
3. Patient under tutorship or guardianship.
4. Dementia, mental alteration or psychiatric pathology influencing patient consent procedure and/or protocol observance and study follow-up.
5. Patient enable to protocol follow-up for psychological, social, familial or geographical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients. | 24 months
  Proportion of patients whose care management was modified at least once and specifically by Moovcare® Lung application at months.
Proportion of patients. | 12 months
  Proportion of patients whose care management was modified at least once and specifically by Moovcare® Lung application at 12 months.

SECONDARY OUTCOMES:
Clinical aspects : date of consultation. | 24 months
  Interval between the date of early consultation or early scan and the date of the scheduled consultation or scan.
Clinical aspects : Number of unscheduled hospitalizations. | 24 months
  Number of unscheduled hospitalizations.
Clinical aspects : Duration of unscheduled hospitalizations. | 24 months
  Duration of unscheduled hospitalizations.
Clinical aspects : Number of overall hospitalizations. | 24 months
  Number of overall hospitalizations.
Clinical aspects : Duration of overall hospitalizations. | 24 months
  Number of overall hospitalizations.
Clinical aspects : Quality of life. | Every 3 months until 24 months
  Quality of life criteria with EORTC QLQ-C30 questionnaire scale.
Clinical aspects : Overall survival over the entire follow-up. | 24 months
  Overall survival over the entire follow-up.
Organizational aspects : number of stakeholders | 24 months
  Number of stakeholders on the application, number of stakeholders specifically recruited for the application and type of stakeholders.
Organizational aspects : Time for each investigating center | 24 months
  Calculation of the time spent to set up the protocol and the application for each investigating center.
Organizational aspects : Functioning and processing of alerts : | 24 months
  Time spent to register patients.
Organizational aspects : Functioning and processing of alerts : | 24 months
  Total number of alerts, rate of alerts handled by the health care team.
Organizational aspects : Functioning and processing of alerts : | 24 months
  Number of alerts that led to an early consultation: processing time, type of provider(s), number of alerts that led to further investigation and the type of investigation: processing time, type of provider(s), rate of alerts that led to a change in management.
Organizational aspects : Functioning and processing of alerts : | 24 months
  Relevant post-alert management time, as well as the number of stakeholders on the application, type of stakeholders.
Organizational aspects : Patient satisfaction. | 3, 6, 12, 18 and 24 months of use of the application
  The degree of patient satisfaction will be evaluated with a satisfaction questionnaire. A form to be filled in after 3, 6, 12, 18 and 24 months of use of the application.
Organizational aspects : Satisfaction of the care teams at 6 months follow-up. | 6 months follow-up
  Physician satisfaction: the satisfaction of all doctors involved will be evaluated with a questionnaire to be filled in (Questionnaire Satisfaction Médecins).
  Staff satisfaction: the satisfaction of all staff involved (coordinating nurses, secretaries or other categories of staff) will be assessed with a questionnaire to be filled in (Questionnaire Satisfaction Collaborateur).
Organizational aspects : Patient compliance. | 24 months
  The compliance will be evaluated by the ratio between the number of completed questionnaires and the invitation's number sent to complete them. Reasons of impossible connection (must be documented on medical records) will be subtracted from the calculation.
  The number of patients who voluntary abandoned the use of Moovcare® Lung medical device will be reduced considered as non-compliant.
Organizational aspects : all secondary outcome measures | 12 months of follow-up
  above criteria will be assessed at 12 months of follow-up. This analysis will be done one year after inclusion of the last patient.

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Chu Argenteuil, Argenteuil
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - Hôpital Forcilles, Férolles-Attilly
  - Hôpital Nord-Ouest, Gleizé
  - Hopital Franco Britannique, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Polyclinique de Limoges - Site de François CHENIEUX, Limoges
  - AP-HM La Timone, Marseille
  - Clinique Saint-George, Nice
  - Institut Curie, Paris
  - CHU de PAU, Pau
  - Institut Curie, Saint-Cloud
  - Clinique mutualiste de l'ESTUAIRE, Saint-Nazaire
  - Nouvel Hôpital Civil, Strasbourg
  - Hopital Robert Schumann, Vantoux

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).